CLINICAL TRIAL: NCT05646199
Title: The Effect of Semaglutide Compared to Metformin in Obese Women With Polycystic Ovary Syndrome (PCOS): a Randomised Controlled Study (Semaglutide-PCOS Trial).
Brief Title: Semaglutide vs Metformin in Polycystic Ovary Syndrome (PCOS)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2603
Record Dates: First submitted 2022-11-17; First posted 2022-12-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Participants in this group will be given metformin
  Interventions: Drug: Metformin
- Semaglutide (Active Comparator): Participants in this group with receive Semaglutide
  Interventions: Drug: Semaglutide Injectable Product

INTERVENTIONS:
Drug: Metformin — Participants will receive metformin
  Arms: Metformin
Drug: Semaglutide Injectable Product — Participants in this group will receive injectable Semaglutide
  Arms: Semaglutide

SUMMARY:
The goal of this clinical trial is to compare the effect of Semaglutide and metformin on weight loss in obese women with Polycystic Ovarian Syndrome (PCOS) over a 28-week treatment period.

The main question it aims to answer is:

• Which of the 2 drugs, metformin or Semaglutide causes more weight loss when used over a 28 week treatment period in obese women with PCOS?

Participants will be divided into 2 groups by chance. In the first group, participants will be asked to take metformin orally. In the second group, participants will take Semaglutide by injection under the skin weekly.

The maximum duration of participation for the patients in the trial is 32 weeks.

Researchers will compare the weight reduction, quality of life and individuals' wellbeing between the two groups.

DETAILED DESCRIPTION:
Background:

Polycystic ovary syndrome (PCOS) is one of the most common metabolic disorders that affects 6-20% of reproductive-aged women and has an increased risk for type 2 diabetes mellitus (T2DM) and cardiovascular disease. Obesity affects more than 50% of women with PCOS and has been demonstrated to play a vital role in the establishment of symptoms in these patients. Bariatric surgery has been shown to improve metabolic parameters but reports of dietary intervention studies have been variable. PCOS is associated with an increased risk of depressive symptoms and a low quality of life (QOL) with weight being a major contributor. Even modest weight loss of 5% of initial body weight has been shown to improve menstrual disturbance, testosterone levels, hyperlipidaemia, and insulin resistance in women with PCOS. Metformin, most commonly used medication for PCOS works by improving insulin sensitivity in peripheral tissues, inhibit hepatic glucose production and increase glucose disposal by the peripheral tissues.

It has been used for decades in treatment of PCOS with improvement in menstrual irregularities and possible reduction of androgen levels. However, the effect of metformin on body weight (a major contributor of pathophysiology and symptoms in PCOS) remained highly variable between these patients. The first observational study of metformin in PCOS reported weight loss during metformin therapy. In a randomised controlled trial (RCT) designed to investigate the effect of metformin in body weight reported a significant decrease in BMI in obese women independent of their lifestyle. The recent meta-analysis assessed the effectiveness of metformin in PCOS reported a significant effect on body mass index (BMI) in women with PCOS. It is clear, however, that metformin does not increase body weight and might help to limit weight gain. Along with wide variation in response metformin is not tolerated by 10-20% of women with PCOS mainly due to its gastrointestinal side effects. Therefore, it is imperative that investigators look beyond metformin in obese women with PCOS, as this has shown to improve metabolic and hormonal parameters.

In a pilot study, another glucagon like peptide - 1 receptor agonist (GLP-1RA), liraglutide 1.8mg daily for 6 months reduced weight in obese women with PCOS and age and body mass index matched control women. They also demonstrated that liraglutide 1.8mg daily for 6 months in young obese women with PCOS showed significant improvement in physical health, social health, psychological and hence quality of life in this group.

Semaglutide a new GLP-1RA approved as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes and is associated with significant weight loss. In patients with type 2 diabetes, there was ≥5% weight loss in 63% of patients treated with Semaglutide. On the other hand, liraglutide has shown around 5-7 kg of weight reduction from the baseline in patient with T2DM. However, it has been previously reported in the SUSTAIN trials, Semaglutide-treated subjects have achieved a significant weight loss of >10% compared to placebo. The effect of Semaglutide on weight loss and resultant improvement in the metabolic parameters and QOL in women with PCOS is unknown. In a recent double-blind randomized trial, compared Semaglutide to liraglutide in obese patients with no diabetes has shown a significant weight loss compared to placebo. Liraglutide is administered as a daily subcutaneous injection whereas Semaglutide is administered as a weekly subcutaneous injection. Therefore, investigators are conducting this trial to assess the feasibility and trying to replicate the greater weight loss with Semaglutide that has already been shown in other trial, in obese women with PCOS.

Overall hypothesis:

Treatment with Semaglutide will result in significant weight loss compared to metformin and that will be associated with significant improvements in hormonal and metabolic parameters, quality of life and cardiovascular risk factors as secondary endpoints in obese women with PCOS.

This is a randomized controlled trial

The trial consists of 7 visits and 3 telephone calls. Patients will be randomized on a 1:1 ratio to receive either:

Semaglutide 0.25mg subcutaneous weekly for 4 weeks followed by semaglutide 0.5 mg weekly for 4 weeks, then escalating to semaglutide 1 mg/ week for 4 weeks, followed by semaglutide 1.7 mg/week for 4 weeks before titrated up to maximum dose of 2.4 mg a week for 12 weeks if tolerated.

Or Metformin 500 mg/ day for 1 week followed by 500mg/twice a day for 1 week titrated up to 500 mg / day with breakfast and 1000 mg/ day with evening meals for 26 weeks if tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide signed informed consent prior to any trial activity.
2. Women, aged 18-45 years (inclusive), with confirmed diagnosis of PCOS based on Rotterdam criteria [12].
3. Body mass index ≥30 kg/m2
4. Negative pregnancy test during screening visit and agree to use barrier contraception during the study period.
5. Participants from all ethnicities who are English speakers

Exclusion Criteria:

1. Non-classical 21-hydroxylase deficiency, hyperprolactinaemia, Cushing's disease, and androgen-secreting tumours will be excluded by appropriate tests.
2. Confirmed type 2 diabetes and type 1 diabetes.
3. Pregnancy, breastfeeding or intends to become pregnant.
4. Subjects who are on any of the following medications within 3 months of screening:

   * Metformin or other insulin-sensitizing medications (e.g. pioglitazone)
   * Hormonal contraceptives (e.g. birth control pills, hormone-releasing implants. Locally acting hormone - containing IUD such as Mirena coil is permitted).
   * Anti-androgens (e.g., spironolactone, flutamide, finasteride, etc.)
   * Clomiphene citrate or oestrogen modulators such as letrozole
   * GnRH modulators such as leuprolide
   * Minoxidil
5. Have been involved in another medicinal trial (CTIMP) within the past four weeks.
6. Presence or history of neoplasm within 5 years prior to screening. Basal skin carcinoma is allowed.
7. History of pancreatitis
8. Any regular medications that would affect weight management (such as steroids)
9. Any contraindications for treatment with semaglutide.
10. Participants under 18 years
11. Participants who cannot adequately understand verbal and / or written explanations given in English.
12. Confirmed excessive and compulsive drinking of alcohol i.e., alcohol abuse as determined from GP medical notes by the Fast Alcohol Screening Test (FAST) or history of previous alcohol abuse.
13. Moderate to severe renal impairment (creatinine clearance [CrCl] ≤ 60 ml/min or estimated glomerular filtration rate [eGFR] ≤ 60 ml/min/1.73 m2.
14. Severe hepatic insufficiency / and or significant abnormal liver function defines as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and / or alanine aminotransferase (ALT) > 3ULN.
15. History of a major surgical procedure involving the stomach or small intestine which could affect absorption as judged by the investigator.
16. Have severe and enduring mental health problems.
17. Personal or first-degree relative history of multiple endocrine neoplasia type 2 (MEN2) or medullary thyroid cancer (MTC).
18. Clinical or radiological evidence of thyroid nodules.
19. Any contraindication to the administration of metformin.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Weight loss (kg) | 28 weeks
  Changes in weight from baseline

SECONDARY OUTCOMES:
Fat mass | 28 weeks
  Changes in body fat percentage (%) measured using TANITA
Free androgen index (FAI) | 28 weeks
  Changes in Free androgen index (%) calculated from testosterone and sex hormone binding globulin; FAI= (Total Testosterone/Sex Hormone binding globulin)X100%
Blood pressure | 28 weeks
  Changes in blood pressure (mmHg)
Pulse rate | 28 weeks
  Changes in pulse rate (beats per minute)
Glucose tolerance | 28 weeks
  Changes in glucose reading (mmol/l) at 2 hours following 75g of oral glucose

CONTACTS AND LOCATIONS:
Overall Officials: Thozhukat Sathyapalan, MD, FRCP, Principal Investigator — University of Hull
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teede HJ, Joham AE, Paul E, Moran LJ, Loxton D, Jolley D, Lombard C. Longitudinal weight gain in women identified with polycystic ovary syndrome: results of an observational study in young women. Obesity (Silver Spring). 2013 Aug;21(8):1526-32. doi: 10.1002/oby.20213. Epub 2013 Jul 2. PMID 23818329
- [Background] Ovalle F, Azziz R. Insulin resistance, polycystic ovary syndrome, and type 2 diabetes mellitus. Fertil Steril. 2002 Jun;77(6):1095-105. doi: 10.1016/s0015-0282(02)03111-4. PMID 12057712
- [Background] Shaw LJ, Bairey Merz CN, Azziz R, Stanczyk FZ, Sopko G, Braunstein GD, Kelsey SF, Kip KE, Cooper-Dehoff RM, Johnson BD, Vaccarino V, Reis SE, Bittner V, Hodgson TK, Rogers W, Pepine CJ. Postmenopausal women with a history of irregular menses and elevated androgen measurements at high risk for worsening cardiovascular event-free survival: results from the National Institutes of Health--National Heart, Lung, and Blood Institute sponsored Women's Ischemia Syndrome Evaluation. J Clin Endocrinol Metab. 2008 Apr;93(4):1276-84. doi: 10.1210/jc.2007-0425. Epub 2008 Jan 8. PMID 18182456 (Retraction: PMID 25701302 J Clin Endocrinol Metab. 2015 Mar;100(3):1206)
- [Background] Yildiz BO, Knochenhauer ES, Azziz R. Impact of obesity on the risk for polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Jan;93(1):162-8. doi: 10.1210/jc.2007-1834. Epub 2007 Oct 9. PMID 17925334
- [Background] Skubleny D, Switzer NJ, Gill RS, Dykstra M, Shi X, Sagle MA, de Gara C, Birch DW, Karmali S. The Impact of Bariatric Surgery on Polycystic Ovary Syndrome: a Systematic Review and Meta-analysis. Obes Surg. 2016 Jan;26(1):169-76. doi: 10.1007/s11695-015-1902-5. PMID 26431698
- [Background] Moran LJ, Ko H, Misso M, Marsh K, Noakes M, Talbot M, Frearson M, Thondan M, Stepto N, Teede HJ. Dietary composition in the treatment of polycystic ovary syndrome: a systematic review to inform evidence-based guidelines. Hum Reprod Update. 2013 Sep-Oct;19(5):432. doi: 10.1093/humupd/dmt015. Epub 2013 May 31. No abstract available. PMID 23727939
- [Background] Thomson RL, Brinkworth GD, Noakes M, Clifton PM, Norman RJ, Buckley JD. The effect of diet and exercise on markers of endothelial function in overweight and obese women with polycystic ovary syndrome. Hum Reprod. 2012 Jul;27(7):2169-76. doi: 10.1093/humrep/des138. Epub 2012 May 2. PMID 22552687
- [Background] Barnard L, Ferriday D, Guenther N, Strauss B, Balen AH, Dye L. Quality of life and psychological well being in polycystic ovary syndrome. Hum Reprod. 2007 Aug;22(8):2279-86. doi: 10.1093/humrep/dem108. Epub 2007 May 30. PMID 17537782
- [Background] Thomson RL, Buckley JD, Noakes M, Clifton PM, Norman RJ, Brinkworth GD. The effect of a hypocaloric diet with and without exercise training on body composition, cardiometabolic risk profile, and reproductive function in overweight and obese women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Sep;93(9):3373-80. doi: 10.1210/jc.2008-0751. Epub 2008 Jun 26. PMID 18583464
- [Background] Sathyapalan T, Cho LW, Kilpatrick ES, Coady AM, Atkin SL. A comparison between rimonabant and metformin in reducing biochemical hyperandrogenaemia and insulin resistance in patients with polycystic ovary syndrome (PCOS): a randomized open-label parallel study. Clin Endocrinol (Oxf). 2008 Dec;69(6):931-5. doi: 10.1111/j.1365-2265.2008.03260.x. Epub 2008 Apr 10. PMID 18410553